CLINICAL TRIAL: NCT03465735
Title: Efficacy and Safety of Vascular Boot Warming Program After Acute DVT±PE for Earlier Resolution of Venous Thromboembolism (VTE) and Prevention of Post Thrombotic Syndrome: A Pilot Study.
Brief Title: Vascular Boot Warming Program After Acute Deep Vein Thrombosis (DVT) ± Pulmonary Embolism (PE)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of recruitment of eligible participants
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Waldemar E. Wysokinski, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-008129
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-05

CONDITIONS: Acute DVT of Lower Extremity
Keywords: Deep; Pulmonary; Venous; Vascular; Post; Vein; Thrombosis; Embolism; Thromboembolism; Thrombotic; Syndrome
MeSH Terms: conditions — Thrombosis; Embolism; Thromboembolism; Syndrome | interventions — Standard of Care; Heparin; Enoxaparin; Dalteparin; Warfarin; Vitamin B 6; Dabigatran; Rivaroxaban; apixaban; edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Other): Ultrasound of the leg with DVT and leg circumference measurement at 3 days, 10 days, and 3 months. Ultrasound data will include data on thrombus resolution, such as size and recanalization present.
  Interventions: Drug: Standard of Care
- Vascular Boot Group (Other): For each vascular boot session, the following data will be recorded:
  Wearing the vascular boot during first 10 days of study for minimum of 30 minutes per day
  Interventions: Combination Product: Vascular Boot; Drug: Standard of Care

INTERVENTIONS:
Combination Product: Vascular Boot — The Vascular Boot is one size fits all, insulated fleece padding, and cell foam to enhance and maintain lower limb warmth while maintaining no pressure points on the lower extremity.
  Other Names: Rooke Boot
  Arms: Vascular Boot Group
Drug: Standard of Care — Anticoagulant therapy will be decided by physician and patient.
  Other Names: Heparin; Enoxaparin (Lovenox); Dalteparin (Fragmin); Warfarin (Coumadin, Jantoven); Dabigatran (Pradaxa); Rivaroxaban (Xarelto); Apixaban (Eliquis); Edoxaban (Savaysa)

SUMMARY:
The Researchers are studying whether a vascular boot warming program plus standard of care anticoagulation can be a safe and effective method to resolve Deep Vein Thrombosis (DVT) ±Pulmonary Embolism (PE) earlier and prevent development of post-thrombotic syndrome (PTS). Additionally, to learn whether a more detailed imaging of the affected lower extremities will provide a more accurate and reliable method to guide treatment for this condition.

DETAILED DESCRIPTION:
Participants with diagnosis of acute lower extremity DVT (proximal and distal) and/or pulmonary embolism will be identified and approached for participation, when they are seen in the Thrombophilia Clinic or Mayo Hospital for management of the acute VTE. If they match the preset inclusion and exclusion criteria, they would then be consented during this visit and scheduled for baseline studies at a later date. Baseline tests include Venous plethysmorgraphy, Lower Extremity Ultrasound, and Medical history, will be conducted and if eligible, participant will then be randomized to vascular boot plus standard anti coagulation program or standard anti coagulation using a randomization program. Participants will be randomized into two groups and followed for 3 months. Standard of Care (SOC) Group (no vascular boot utilized): Patients will receive standard anticoagulation (determined at discretion of the treating provider), baseline studies, and follow up at the end of treatment (3months). Vascular Boot (VB) Group (includes vascular boot in addition to SOC): Patients will receive standard anticoagulation (determined at discretion of the treating provider), baseline studies and standardized vascular boot warming. All patients randomized to this group will wear the vascular boot for a minimum of 30 minutes per day for the first 10 days of participation. Patients in this group may initially be enrolled at either the thrombophilia clinic or the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Able to tolerate wearing a vascular boot, if randomized to this group.
* Diagnosis of acute DVT±PE (within 24 - 48 hours) and received approximately 24 hours of anticoagulation prior to starting the study.

Exclusion Criteria:

* Unable to tolerate wearing a vascular boot
* Unable to comply with keeping log of activity/ of wearing a vascular boot.
* Weight > 300 pounds. (weight limit for the venous plethysmography chair)
* Previous history of DVT or PE.
* On anticoagulation for another purpose (example stroke prevention with atrial fibrillation).
* Patients who do not accept to participate in research studies.
* Pregnant women will not be allowed to participate
* Patients less than 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2020-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar E Wysokinski, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heit JA. The epidemiology of venous thromboembolism in the community. Arterioscler Thromb Vasc Biol. 2008 Mar;28(3):370-2. doi: 10.1161/ATVBAHA.108.162545. No abstract available. PMID 18296591
- [Background] Centers for Disease Control and Prevention (CDC). Venous thromboembolism in adult hospitalizations - United States, 2007-2009. MMWR Morb Mortal Wkly Rep. 2012 Jun 8;61(22):401-4. PMID 22672974
- [Background] Heit JA, Crusan DJ, Ashrani AA, Petterson TM, Bailey KR. Venous thromboembolism attack rates among recently hospitalized vs. community residents: a population-based cohort study. JAMA. 2015 in submission.
- [Background] Heit JA, Ashrani AA, Crusan DJ, Petterson TM, Bailey KR. Trends in venous thromboembolism incidence, 1981-2010: a population-based cohort study. JAMA. 2015, in submission.
- [Background] Kahn SR, Comerota AJ, Cushman M, Evans NS, Ginsberg JS, Goldenberg NA, Gupta DK, Prandoni P, Vedantham S, Walsh ME, Weitz JI; American Heart Association Council on Peripheral Vascular Disease, Council on Clinical Cardiology, and Council on Cardiovascular and Stroke Nursing. The postthrombotic syndrome: evidence-based prevention, diagnosis, and treatment strategies: a scientific statement from the American Heart Association. Circulation. 2014 Oct 28;130(18):1636-61. doi: 10.1161/CIR.0000000000000130. Epub 2014 Sep 22. No abstract available. PMID 25246013
- [Background] Kahn SR, Shapiro S, Wells PS, Rodger MA, Kovacs MJ, Anderson DR, Tagalakis V, Houweling AH, Ducruet T, Holcroft C, Johri M, Solymoss S, Miron MJ, Yeo E, Smith R, Schulman S, Kassis J, Kearon C, Chagnon I, Wong T, Demers C, Hanmiah R, Kaatz S, Selby R, Rathbun S, Desmarais S, Opatrny L, Ortel TL, Ginsberg JS; SOX trial investigators. Compression stockings to prevent post-thrombotic syndrome: a randomised placebo-controlled trial. Lancet. 2014 Mar 8;383(9920):880-8. doi: 10.1016/S0140-6736(13)61902-9. Epub 2013 Dec 6. PMID 24315521
- [Background] O'shaughnessy AM, Fitzgerald DE. The patterns and distribution of residual abnormalities between the individual proximal venous segments after an acute deep vein thrombosis. J Vasc Surg. 2001 Feb;33(2):379-84. doi: 10.1067/mva.2001.111983. PMID 11174793
- [Background] Killewich LA, Macko RF, Cox K, Franklin DR, Benjamin ME, Lilly MP, Flinn WR. Regression of proximal deep venous thrombosis is associated with fibrinolytic enhancement. J Vasc Surg. 1997 Nov;26(5):861-8. doi: 10.1016/s0741-5214(97)70101-0. PMID 9372826
- [Background] Killewich LA, Bedford GR, Beach KW, Strandness DE Jr. Spontaneous lysis of deep venous thrombi: rate and outcome. J Vasc Surg. 1989 Jan;9(1):89-97. PMID 2911146
- [Background] van Ramshorst B, van Bemmelen PS, Hoeneveld H, Faber JA, Eikelboom BC. Thrombus regression in deep venous thrombosis. Quantification of spontaneous thrombolysis with duplex scanning. Circulation. 1992 Aug;86(2):414-9. doi: 10.1161/01.cir.86.2.414. PMID 1638710
- [Background] Caprini JA, Arcelus JI, Hoffman KN, Size G, Laubach M, Traverso CI, Coats R, Finke N, Reyna JJ. Venous duplex imaging follow-up of acute symptomatic deep vein thrombosis of the leg. J Vasc Surg. 1995 Mar;21(3):472-6. doi: 10.1016/s0741-5214(95)70289-x. PMID 7877229
- [Background] Meyer G, Vicaut E, Danays T, Agnelli G, Becattini C, Beyer-Westendorf J, Bluhmki E, Bouvaist H, Brenner B, Couturaud F, Dellas C, Empen K, Franca A, Galie N, Geibel A, Goldhaber SZ, Jimenez D, Kozak M, Kupatt C, Kucher N, Lang IM, Lankeit M, Meneveau N, Pacouret G, Palazzini M, Petris A, Pruszczyk P, Rugolotto M, Salvi A, Schellong S, Sebbane M, Sobkowicz B, Stefanovic BS, Thiele H, Torbicki A, Verschuren F, Konstantinides SV; PEITHO Investigators. Fibrinolysis for patients with intermediate-risk pulmonary embolism. N Engl J Med. 2014 Apr 10;370(15):1402-11. doi: 10.1056/NEJMoa1302097. PMID 24716681
- [Background] Piazza G, Hohlfelder B, Jaff MR, Ouriel K, Engelhardt TC, Sterling KM, Jones NJ, Gurley JC, Bhatheja R, Kennedy RJ, Goswami N, Natarajan K, Rundback J, Sadiq IR, Liu SK, Bhalla N, Raja ML, Weinstock BS, Cynamon J, Elmasri FF, Garcia MJ, Kumar M, Ayerdi J, Soukas P, Kuo W, Liu PY, Goldhaber SZ; SEATTLE II Investigators. A Prospective, Single-Arm, Multicenter Trial of Ultrasound-Facilitated, Catheter-Directed, Low-Dose Fibrinolysis for Acute Massive and Submassive Pulmonary Embolism: The SEATTLE II Study. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1382-1392. doi: 10.1016/j.jcin.2015.04.020. PMID 26315743
- [Background] Ogawa T, Hoshino S, Midorikawa H, Sato K. Intermittent pneumatic compression of the foot and calf improves the outcome of catheter-directed thrombolysis using low-dose urokinase in patients with acute proximal venous thrombosis of the leg. J Vasc Surg. 2005 Nov;42(5):940-4. doi: 10.1016/j.jvs.2005.07.041. PMID 16275451
- [Background] Murphy TP, Cutlip DE, Regensteiner JG, Mohler ER, Cohen DJ, Reynolds MR, Massaro JM, Lewis BA, Cerezo J, Oldenburg NC, Thum CC, Goldberg S, Jaff MR, Steffes MW, Comerota AJ, Ehrman J, Treat-Jacobson D, Walsh ME, Collins T, Badenhop DT, Bronas U, Hirsch AT; CLEVER Study Investigators. Supervised exercise versus primary stenting for claudication resulting from aortoiliac peripheral artery disease: six-month outcomes from the claudication: exercise versus endoluminal revascularization (CLEVER) study. Circulation. 2012 Jan 3;125(1):130-9. doi: 10.1161/CIRCULATIONAHA.111.075770. Epub 2011 Nov 16. PMID 22090168
- [Background] Recek C. Calf pump activity influencing venous hemodynamics in the lower extremity. Int J Angiol. 2013 Mar;22(1):23-30. doi: 10.1055/s-0033-1334092. PMID 24436580
- [Background] Labropoulos N, Giannoukas AD, Nicolaides AN, Veller M, Leon M, Volteas N. The role of venous reflux and calf muscle pump function in nonthrombotic chronic venous insufficiency. Correlation with severity of signs and symptoms. Arch Surg. 1996 Apr;131(4):403-6. doi: 10.1001/archsurg.1996.01430160061011. PMID 8615726
- [Background] Kahn SR, Azoulay L, Hirsch A, Haber M, Strulovitch C, Shrier I. Acute effects of exercise in patients with previous deep venous thrombosis: impact of the postthrombotic syndrome. Chest. 2003 Feb;123(2):399-405. doi: 10.1378/chest.123.2.399. PMID 12576357
- [Background] Shrier I, Kahn SR. Effect of physical activity after recent deep venous thrombosis: a cohort study. Med Sci Sports Exerc. 2005 Apr;37(4):630-4. doi: 10.1249/01.mss.0000158192.07412.89. PMID 15809562
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Vascular Boot Group: For each vascular boot session, the following data will be recorded:
  Wearing the vascular boot during first 10 days of study for minimum of 30 minutes per day
  Vascular Boot: The Vascular Boot is one size fits all, insulated fleece padding, and cell foam to enhance and maintain lower limb warmth while maintaining no pressure points on the lower extremity.
  Standard of Care: Anticoagulant therapy will be decided by physician and patient.
Period: Overall Study
Arm/Group | Standard of Care | Vascular Boot Group
Started | 8 | 7
Completed | 7 | 5
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Vascular Boot Group | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (17.5) | 66.4 (13.6) | 61.1 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 4 | 1 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Affected Leg Pain
Description: Affected leg pain measured on a 0-10 scale. 0 indicating No pain and 10 indicating Worst Possible Pain.
Time Frame: baseline, 10 days
Population: Study terminated due to lack of recruitment of eligible participants. Data was not analyzed due to lack of recruitment. Data not analyzed and no longer available to be analyzed.
Arm/Group | Standard of Care | Vascular Boot Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collect on each subject from baseline to end of anti coagulation program for approximately a total of three months.
Arm/Group | Standard of Care | Vascular Boot Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 7/8 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=8) | Vascular Boot Group (N=7)
Occlusive thrombi (Cardiac disorders) | 1 (1) | 0 (0)
Thoracic Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Chemical Exposure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Left adnexal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to lack of recruitment of eligible participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/35/NCT03465735/Prot_SAP_000.pdf